CLINICAL TRIAL: NCT03703895
Title: "A Double-Blind, Pilot Study to Evaluate the Efficacy and Safety of Topical AFX 5931 in the Treatment of Mild to Moderate Hand Dermatitis"
Brief Title: A Study for a Topical Medication Versus Placebo in Patients With Hand Dermatitis
Acronym: AFX5931
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: Afecta Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCCR 08-2018; AFX5931-A 07312018 (Other: Afecta Pharmaceuticals)
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Results first posted 2022-11-23 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Hand Dermatitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator (Active Comparator): Active Comparator, Topical AFX5931, a medication combining a small, potent anti-inflammatory molecule. Subjects will complete up to 4 study visits where Topical AFX5931 will be applied twice daily for 28 days.
  Interventions: Drug: Topical AFX5931
- Placebo Comparator (Placebo Comparator): Placebo Comparator, Topical Placebo. Subjects will complete up to 4 study visits where Topical Placebo will be applied twice daily for 28 days.
  Interventions: Drug: Topical Placebo

INTERVENTIONS:
Drug: Topical AFX5931 — Active Comparator, Topical AFX5931, a medication combining a small, potent anti-inflammatory molecule.
  Arms: Active Comparator
Drug: Topical Placebo — Placebo Comparator, Topical Placebo.
  Arms: Placebo Comparator

SUMMARY:
This is a double-blind, pilot study with 20 subjects to determine the tolerability and efficacy of topical AFX 5931 in the treatment of mild to moderate hand dermatitis. Subjects are screened up to 30 days before the baseline visit. Subjects who meet the eligibility criteria may qualify for the study. Subjects will be randomized in a 3:1 ratio to receive either the active or vehicle medication. 15 subjects will receive the active, therapeutic product and 5 subjects will receive the inactive, vehicle product.

DETAILED DESCRIPTION:
This is a double-blind, pilot study with 20 subjects to determine the tolerability and efficacy of topical AFX 5931 in the treatment of mild to moderate hand dermatitis. Subjects are screened up to 30 days before the baseline visit. Subjects who meet the eligibility criteria may qualify for the study. Subjects will be randomized in a 3:1 ratio to receive either the active or vehicle medication. 15 subjects will receive the active, therapeutic product and 5 subjects will receive the inactive, vehicle product. Subjects will complete 4 study visits according to the following 4-week timeline: Day [-30] - [-1] (Screening), Day 0 (Baseline), Day 14 (Follow-Up), Day 28 (Follow-up | ET | EOS). At Visit 2, IP will be dispensed and baseline readings of efficacy as well as safety/tolerability assessments will be obtained prior to application of the IP. Subjects will apply IP twice daily and compliance will be monitored by periodically reviewing the subject diary. The evaluations that will be used to measure efficacy of the product will be the Investigator's Global Assessment and Hand Eczema Severity Index. The Subject's Local Dermal Tolerability Assessment and Local Skin Reaction Assessment will be used throughout the course of the study to evaluate tolerability. Additionally, the actions that will be taken to evaluate safety will be the monitoring of adverse events, vital signs, and changes in concomitant medications. Digital photographs will be taken at each visit (excluding Visit 3).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or non-pregnant female, 12 years of age and older.
2. Subject is willing and able to provide written informed consent for the study.
3. Subject is willing and able to apply the investigational product as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
4. Subject has clinical diagnosis of mild to moderate hand dermatitis for at least 3 months.
5. Subject has a baseline Investigator's Global Assessment (IGA) score of 2 or 3 (disease severity of mild or moderate).
6. Subject is in good general health and free of any disease state or physical condition that might impair evaluation of hand dermatitis or which, in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.
7. Women of childbearing potential (WOCBP) must use an effective method of birth control or must be post-menopausal or surgically sterile. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Baseline.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject is currently enrolled in an investigational drug or device study.
3. Subject has used an investigational drug or investigational device treatment within 30 days prior to Visit 2/Baseline.
4. Subject has active cutaneous bacterial or viral infection in any treatment area (clinically infected hand dermatitis) at Visit 2/Baseline.
5. Subject has used any of the following therapies within 30 days prior to Visit 2/Baseline:

   * Systemic corticosteroids (oral and injectable [intravenous and intramuscular]) (Intranasal and Inhalational steroids are allowed if use is kept constant during the study)
   * UVA/UVB therapy
   * PUVA (psoralen plus ultraviolet A) therapy
   * Immunomodulators or immunosuppressive therapies
   * Interferon
   * Cytotoxic drugs (e.g., methotrexate, cyclophosphamide, azathioprine)
   * Oral retinoids
6. Subject has used any of the following therapies within 14 days prior to Visit 2/Baseline:

   * Systemic antibiotics
   * Topical calcipotriene or other topical vitamin D preparations
7. Subject has used any of the following therapies within 7 days prior to Visit 2/Baseline: • Topical and oral antihistamines

   * Topical antibiotics
   * Topical corticosteroids
   * Topical antifungals
8. Subject has a history of sensitivity to any of the ingredients in the investigational product
9. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, M.D, Ph.D., Principal Investigator — The Center for Clinical and Cosmetic Research
Locations (1):
- The Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Afecta Pharmaceuticals — http://www.afectapharm.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical AFX5931 (Active Comparator): Active Comparator, Topical AFX5931, a medication combining a small, potent anti-inflammatory molecule. 15 healthy male or non pregnant female subjects over the age of 18 will complete up to 4 study visits where Topical AFX5931 will be applied twice daily for 28 days.
  Topical AFX5931: Active Comparator, Topical AFX5931, a medication combining a small, potent anti-inflammatory molecule.
- Placebo Comparator: Placebo Comparator, Topical Placebo. 5 healthy male or non pregnant female subjects over the age of 18 will complete up to 4 study visits where Topical Placebo will be applied twice daily for 28 days.
  Topical Placebo: Placebo Comparator, Topical Placebo.
Period: Overall Study
Arm/Group | Topical AFX5931 (Active Comparator) | Placebo Comparator
Started | 15 | 5
Completed | 15 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Placebo Comparator | Total
Number analyzed (Participants) | 15 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 6 | 0 | 6
Age, Continuous [Mean (Full Range); unit: years] | 55.2 [24 to 58] | 47.8 [18 to 82] | 53.65 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 12 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 10 | 4 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure for Efficacy (IGA)
Description: To measure the efficacy of topical AFX 5931 in the treatment of mild to moderate hand dermatitis in subjects 12 years of age or older assessed via the Investigator's Global Assessment
  The investigator will rate the subject's hand dermatitis on a visual 5-point scale as follows:
  0: Clear: No signs of HE
  1. Almost clear: Just perceptible scaling and/or erythema;
  2. Mild disease: Mild scaling and/or mild erythema, and/or mild cracking
  3. Moderate disease: Moderate scaling and/or erythema, and/or moderate cracking/fissuring
  4. Severe disease: Severe scaling and/or severe erythema, and/or severe cracking/fissuring
  Dorsal and palmar surfaces of the hand are evaluated together.
Time Frame: Baseline; Day 14; Day 28
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 15 | 5
score on a scale
  Baseline | 2.33 [2.09 to 2.57] | 2.20 [1.85 to 2.55]
  Day 14 | 2.43 [2.18 to 2.68] | 2 [2 to 2]
  Day 28 | 2.20 [1.87 to 2.53] | 2.25 [1.87 to 2.63]

2. Primary Outcome: Primary Outcome Measure for Efficacy (HECSI)
Description: To measure the efficacy of topical AFX 5931 in the treatment of mild to moderate hand dermatitis in subjects 12 years of age or older, assessed via the Hand Eczema Severity Index (HECSI).
  * Investigator-rated clinical evaluation
  * Locations: fingertips, fingers (excluding tips), palms of hands, backs of hands, wrists
  * Intensity: graded on a visual 4-point scale (0 = no skin changes, 1 = mild disease, 2 = moderate, 3 = severe) for each Clinical sign (erythema, infiltration/papulation, vesicles, figures, scaling, and edema) at each location.
  * Extent: graded on a visual 5-point scale (0 = 0% ; 1 = 1-25% ; 2 = 26-50% ; 3 = 51-75% ; 4 = 76-100%) for each location.
  * Total HECSI score (0 to a maximum severity score of 360): the sum of the Intensity of clinical signs multiplied by the Extent grade for each location. The sum of the location scores is the Total HECSI score.
Time Frame: Baseline; Day 14; Day 28
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 15 | 5
units on a scale
  Baseline | 22.67 [19.92 to 25.41] | 25.6 [22.74 to 28.46]
  Day 14 | 20.8 [17.17 to 24.43] | 20 [17.23 to 22.77]
  Day 28 | 20.6 [16.33 to 24.87] | 21 [15.54 to 26.46]

3. Secondary Outcome: Secondary Outcome Measures for Tolerability and Safety (Tolerability Assessment - Pruritus Score)
Description: The subjects will be asked to grade their feeling of itching at the application site using a 4-point tolerability scale, where 0=None, 1= Mild, 2= Moderate, and 3=Severe.
  Pruritus: Definition: itching 0 = None: No itching
  1. = Mild: Occasional, slight itching/scratching
  2. = Moderate: Constant or intermittent itching/scratching/discomfort that is not disturbing sleep
  3. = Severe: Bothersome itching/scratching/discomfort that is disturbing sleep
Time Frame: Baseline; Day 14; Day 28
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 15 | 5
units on a scale
  Baseline | 1.53 [1.28 to 1.79] | 1.8 [1.14 to 2.46]
  Day 14 | 1.29 [0.80 to 1.77] | 1 [0.22 to 1.78]
  Day 28 | 0.93 [0.50 to 1.37] | 1 [0.38 to 1.62]

4. Secondary Outcome: Secondary Outcome Measures for Tolerability and Safety (LSR)
Description: The investigator/ designee will describe their Local Skin Reaction (LSR) assessment of the subject's hands using a 4-point tolerability scale.
  Erythema: abnormal redness of the skin 0 = No erythema
  1. = Mild (Slight pinkness present)
  2. = Moderate (Definite, dull redness that is clearly distinguishable)
  3. = Severe (Intense, deep redness)
  Induration/Papulation: inflammation, swelling 0 = No elevation
  1. = Mild (Slightly perceptible elevation)
  2. = Moderate (Clearly perceptible elevation but not extensive)
  3. = Severe (Marked and extensive elevation)
  Lichenification: thickening upper layers of skin 0 = No thickening
  1. = Mild (Slight thickening of skin discernible only by touch and with skin markings minimally exaggerated)
  2. = Moderate (Definite thickening of the skin with skin markings exaggerated so that they form a visible crisscross pattern)
  3. = Severe (Thickened, indurated skin with skin markings visibly portraying an exaggerated crisscross pattern)
Time Frame: Baseline; Day 14; Day 28
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Comparator | Placebo Comparator
Number analyzed (Participants) | 15 | 5
units on a scale
  Baseline (Erythema) | 1.33 [1.09 to 1.57] | 1.4 [0.97 to 1.83]
  Day 14 (Erythema) | 1.36 [1.11 to 1.60] | 1 [1 to 1]
  Day 28 (Erythema) | 1.27 [1.04 to 1.49] | 1.25 [0.87 to 1.63]
  Baseline (Induration) | 1.27 [1.04 to 1.49] | 1.2 [0.85 to 1.55]
  Day 14 (Induration) | 1.21 [1.01 to 1.42] | 1 [1 to 1]
  Day 28 (Induration) | 1.2 [0.87 to 1.53] | 1.25 [0.87 to 1.63]
  Baseline (Lichenification) | 1.47 [1.21 to 1.72] | 1.8 [1.45 to 2.15]
  Day 14 (Lichenification) | 1.57 [1.26 to 1.89] | 1.4 [0.97 to 1.83]
  Day 28 (Lichenification) | 1.4 [1.15 to 1.65] | 1.5 [1.06 to 1.94]

5. Secondary Outcome: Measures for Safety (Adverse Events/Concomitant Medications)
Description: Monitoring the record of AEs (Adverse Events) and changes in concomitant medication/ procedures throughout the course of the study will be the primary mode of safety evaluation.
  At each level of summarization (global, body system, and preferred term), a subject will be counted once if they reported one or more AEs at that level.
  No statistical testing will be performed.
Time Frame: Baseline; Day 14; Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Topical AFX5931 (Active Comparator) | Placebo Comparator
Number analyzed (Participants) | 15 | 5
Participants
  Baseline- Record of AEs | 0 | 0
  Baseline- Changes in concomitant medication/ procedures | 0 | 0
  Day 14- Record of AEs | 0 | 0
  Day 14- Changes in concomitant medication/ procedures | 0 | 0
  Day 28- Record of AEs | 0 | 0
  Day 28- Changes in concomitant medication/ procedures | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Active Comparator | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03703895/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03703895/ICF_002.pdf